CLINICAL TRIAL: NCT03063476
Title: The Effect of Acute Lysine Administration on α-aminoadipic Acid
Brief Title: The Effect of Acute Lysine Administration on α-aminoadipic Acid (Sub-study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jane Ferguson, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 160520-1
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Results first posted 2018-11-30 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy (Experimental): Two healthy subjects will be enrolled and each will undergo study procedures at one visit. After screening and consent have been conducted over the phone, subjects will participate in the study procedures. Subjects will arrive in a fasting state (no eat or drink for 8 hours, excluding water). Following collection of blood pressure, height, weight, and a urine and blood sample, subjects will be given an oral bolus of C-13 labeled lysine (5 g) in 50 ml water. This amount of lysine is equivalent to that which is found in a 5oz. serving of beef. Subjects will provide additional urine and blood samples serially post-ingestion. Because blood draws will be collected through an IV, Normal (0.9%) Saline (NS) will be infused at a rate of approximately 10 ml/hr to flush the canula prior to each blood draw.
  All subjects will undergo the same procedures and interventions.
  Interventions: Drug: C-13 labeled Lysine; Drug: Normal saline

INTERVENTIONS:
Drug: C-13 labeled Lysine — Carbon-13 is a stable naturally occurring heavy isotope of carbon. Inclusion of a 13C label on lysine allows for subsequent differentiation between endogenous and exogenous lysine and 2-AAA for calculation of clearance and excretion of the lysine bolus.
Drug: Normal saline — Because patients will have multiple blood draws during the course of the study, subjects will have an IV placed to reduce the number of needle sticks. To keep the vein open for blood collections, we will infuse Normal (0.9%) Saline (NS) at a rate of approximately 10ml/hr in order to keep the line open.
  Other Names: Normal (0.9%) Saline (NS)

SUMMARY:
This sub-study aims to assess the effect and breakdown of lysine administration, specifically examining whether it leads to increased plasma 2-AAA in healthy humans.

DETAILED DESCRIPTION:
The significance of diabetes and related co-morbidities as considerable health concerns in the US and worldwide is clearly supported by the high incidence (estimated 9.3% of the US population), mortality burden (7th leading cause of death in the US), and rising costs ($245 billion/year). Strategies to identify individuals at high diabetic risk, and to modulate disease processes in these individuals before the onset of overt disease, would have a significant impact in reducing mortality, morbidity and healthcare costs. For this approach to be successful, early markers of disease that predict at-risk individuals before onset of dysregulated glycemic control are required, as well as discovering novel pathways for therapeutic targeting.

The purpose of the study is to investigate a novel biomarker, α-aminoadipic acid (2-AAA), which may influence the risk of diabetes. 2-AAA has been identified as a novel predictor of diabetes development in humans, identifying at-risk individuals before any detectable glucose abnormalities. 2-AAA is a naturally occurring metabolite in the body, and it has no known adverse effects at normal physiological levels. 2-AAA is generated in the body from the breakdown of lysine. Lysine is one of the twenty essential amino acids, meaning that it is essential for human function, but that our body cannot manufacture it. Thus, it is acquired from dietary sources (such as meat, eggs, soybeans and legumes), with a recommended daily intake of 30 mg/kg/day. Amino acids are the building blocks of proteins, which are what allow our cells, organs and body to maintain structure and function. The investigators are interested in whether 2-AAA is increased in the body after consumption of lysine.

The investigators' specific aim is to determine whether acute lysine administration leads to increased plasma 2-AAA in humans. Catabolism of lysine leads to generation of 2-AAA. In this study, the investigators will determine whether a single dose of 13C isotope labeled lysine leads to increased plasma 2-AAA present in the blood and urine of humans. In this sub-study, the investigators will ask 2 lean, healthy subjects (preferably individuals who participated in a previous study visit) to drink a beverage containing C-13 labeled lysine and the investigators will measure the level of 2-AAA in their blood plasma and urine at baseline (before ingestion) and serially post-ingestion. The amount of lysine subjects will be given is equivalent to that which is found in a 5 oz. serving of beef. This sub-study will allow us to further establish and understand the relationship between lysine and 2-AAA in healthy subjects, and inform future studies on how to study the effects of 2-AAA on diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 to <25 kg/m2
* Men and women ages 18-45 years

Exclusion Criteria:

* Current use of prescription medications (apart from hormonal birth control)
* Current use of amino acid supplements (including branched-chain amino acids) or supplemental protein (habitual consumption of protein powder, bars, shakes), and unwilling to temporarily discontinue use (1 week prior to study visit)
* Individuals who currently use tobacco products or have done so in the previous 30 days
* Prior or current cardiovascular disease, renal disease, or liver disease
* Diabetes mellitus (taking insulin, other anti-diabetic agents, or diet-controlled)
* Atrial fibrillation
* Bleeding disorder or anemia
* Positive pregnancy test
* Women who are breastfeeding
* Participation in another clinical trial within the previous 6 weeks prior to the study visit
* Inability to provide written informed consent
* Inability to fast for 8 hours

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane F Ferguson, PhD, Principal Investigator — Vanderbilt Cardiovascular Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects (N=2) were recruited in March 2017. Subjects who had previously participated in a pilot study were invited to return for an additional study visit.
Groups:
- Healthy: Two healthy subjects will be enrolled and each will undergo the same study procedures at one visit.
Period: Overall Study
Arm/Group | Healthy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma 2-AAA Concentration Percentage Change From Baseline
Description: Alpha aminoadipic acid (2-AAA) concentration determined through mass spectrometry, quantified relative to standard.
Time Frame: Baseline and 2-6 hours
Population: Two healthy subjects (one male, one female; one black, one white) were enrolled and completed the study visit.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Healthy
Number analyzed (Participants) | 2
Percentage Change | 63.4 (55)

2. Secondary Outcome: Peak Urinary 2-AAA Concentration Percentage Change From Baseline
Description: Alpha aminoadipic acid (2-AAA) concentration determined through mass spectrometry, quantified relative to standard.
Time Frame: Baseline and 2-6 hours
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Healthy
Number analyzed (Participants) | 2
Percentage change | 39 (99)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 0-6 hours during the study visit.
Arm/Group | Healthy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy (N=2)
Mild Nausea (Gastrointestinal disorders) | 1 (1) — mild wave of nausea onset immediately after drinking solution, subsided within 5 minutes. Subject has not experienced any lingering symptoms or GI distress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03063476/Prot_SAP_000.pdf